CLINICAL TRIAL: NCT05532358
Title: An Open-Label, One-Sequence, Two-Part Drug-Drug Interaction Study in Healthy Volunteers to Assess the CYP1A2 and CYP3A4 Perpetrator Interaction Potential and CYP1A2 Victim Potential of TEV-56286 (anle138b)
Brief Title: A Drug-Drug Interaction Study to Assess the CYP1A2 and CYP3A4 Interaction Potential of TEV-56286 (anle138b)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MODAG GmbH (Industry)
Collaborators: Aptuit (Industry); Quotient Sciences (Industry); Teva Pharmaceutical Industries, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: anle138b-P1-03; 2022-002467-30 (EudraCT Number)
Record Dates: First submitted 2022-09-04; First posted 2022-09-08 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Healthy Volunteers
Keywords: anle138b (TEV-56286); alpha-Synuclein; Oligomer modulator; Multiple System Atrophy; Parkinson Disease; Alzheimer Disease; Neurodegenerative diseases; Tauopathies; Amyloid; Drug-drug interaction
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body; Multiple System Atrophy; Parkinson Disease; Alzheimer Disease; Neurodegenerative Diseases; Tauopathies | interventions — 3-(1,3-benzodioxol-5-yl)-5-(3-bromophenyl)-1H-pyrazole; Caffeine; Midazolam; Fluvoxamine

STUDY DESIGN:
Intervention Model Description: Drug drug interaction study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anle138b (TEV-56286) as perpetrator (part I) (Experimental): Drug: TEV-56286 300 mg QD (single dose and multiple dose for 14 days)
  Victim drugs:
  Caffeine 200 mg Midazolam 2 mg
  Interventions: Drug: anle138b (TEV-56286)
- anle138b (TEV-56286) as victim (part II) (Experimental): Drug: fluvoxamine 100 mg QD for 5 days
  Victim drug:
  TEV-56286 150 mg QD for 14 days + 5 days of co-administation with fluvoxamine
  Interventions: Drug: Fluvoxamine 100 mg QD for 5 days

INTERVENTIONS:
Drug: anle138b (TEV-56286) — Anle138b (TEV-56286) as perpetrator
  Other Names: Caffeine; Midazolam; Fluvoxamine
  Arms: anle138b (TEV-56286) as perpetrator (part I)
Drug: Fluvoxamine 100 mg QD for 5 days — Anle138b (TEV-56286) as victim
  Other Names: TEV-56286 150 mg QD for 14 days + 5 days of co-administation with fluvoxamine
  Arms: anle138b (TEV-56286) as victim (part II)

SUMMARY:
The purpose of this healthy volunteers drug-drug interaction study is to assess the CYP1A2 and CYP3A4 perpetrator interaction potential and CYP1A2 victim potential of TEV-56286 (anle138b).

DETAILED DESCRIPTION:
This a 2-part DDI study that will assess the CYP1A2 and CYP3A4 perpetrator interaction potential of TEV-56286 single dose and multiple dose, using caffeine and midazolam as substrates and CYP1A2 victim potential of TEV-56286 (anle138b) at steady state induction using fluvoxamine as inhibitor [1,2].The estimated time from screening until the follow-up visit is approximately up to 8 weeks for each subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or healthy females of non-childbearing potential
* Must provide written informed consent for participation in the study and must be able to understand the study requirements
* Body mass index (BMI) 18.5 to 32.0 kg/m2.
* Must agree to adhere to the contraception requirements defined in the study protocol.

Exclusion Criteria:

* Serious adverse reaction or serious hypersensitivity to any drug or formulation excipients e.g. fluvoxamine, caffeine, midazolam or benzodiazepines or any of its excipients, or a known drug hypersensitivity idiosyncratic reaction to TEV-56286, or one of its excipients
* History of clinically significant cardiovascular, renal, hepatic, dermatological, chronic respiratory or gastrointestinal disease, neurological or psychiatric disorder, metabolic diseases or a history of any illness that, in the opinion of the investigator, might pose additional risk to the subject by participation in the study or confound the results of the study
* Acute infection and/or antibiotic treatment within 28 days of Day 1
* Major trauma or surgery in the 2 months before screening or at any time between screening and Day 1, or surgery scheduled during the study or follow up period
* History of malignancy or treatment of malignancy in the last 5 years
* History of suicidal ideation with an intent and/or plan and behaviour based upon either clinical history or source documents
* Personal or family history of arrhythmia, sudden unexplained death at a young age (before 40 years) in a first-degree relative, or long QT syndrome, or a personal history of syncope or previous treatment for high blood pressure (BP). Abnormality of 12-lead ECG that may, in the opinion of the investigator, interfere with study participation
* Any procedure or disorder that may interfere with drug absorption, distribution, metabolism, or excretion
* Clinically significant abnormal clinical chemistry, haematology or urinalysis as judged by the investigator.
* Subjects who have received any IMP in a clinical research study within the 90 days prior to Day 1, or less than 5 elimination half-lives prior to Day 1, whichever is longer
* Subjects who are taking, or have taken, any prescribed or over-the-counter drug or herbal remedies in the 14 days before study medication administration or within 5 half-lives whichever is longer.
* Subjects who are taking, or have taken hormonal contraceptives (e.g., oral, patch, injectable or intrauterine device) hormone replacement therapy (HRT) or a long-acting injectable hormonal within 4 weeks prior to first dose of IMP
* Subjects who are taking, or have taken any inducer of CYP 1A2, CYP3A4 within 28 days prior to Day -2
* History of any drug or alcohol abuse in the past 2 years
* Current smokers and those who have smoked within the last 12 months or has a positive urine cotinine test
* Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
* Subjects with a previous history of difficulty in swallowing tablets or capsules, or an anticipated problem with swallowing a large number of capsules
* Subjects who have consumed grapefruit, grapefruit juice, Seville oranges, pomelo-containing products, vegetables from the mustard green family (e.g., kale, broccoli, watercress, collard greens, kohlrabi, brussel sprouts, and mustard) and charbroiled meats within the 14 days prior to Day -2
* Subjects who are unwilling to comply with the restricted use of caffeinated beverages (e.g. coffee, tea, cola) during the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2023-01-28 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Oral pharmacokinetics (PK) of caffeine administered without TEV-56286 in healthy volunteers in the fasted state (Part I). | Day 1
  PK parameter: Cmax for caffeine.
Oral pharmacokinetics (PK) of caffeine administered without TEV-56286 in healthy volunteers in the fasted state (Part I). | Day 1
  PK parameter: AUC(0-inf) for caffeine.
Oral pharmacokinetics (PK) of caffeine administered without TEV-56286 in healthy volunteers in the fasted state (Part I). | Day 1
  PK parameter: AUC (0-last) for caffeine.
Oral pharmacokinetics (PK) of midazolam administered without TEV-56286 in healthy volunteers in the fasted state (Part I). | Day 1
  PK parameter: Cmax for midazolam.
Oral pharmacokinetics (PK) of midazolam administered without TEV-56286 in healthy volunteers in the fasted state (Part I). | Day 1
  PK parameter: AUC(0-inf) for midazolam.
Oral pharmacokinetics (PK) of midazolam administered without TEV-56286 in healthy volunteers in the fasted state (Part I). | Day 1
  PK parameter: AUC (0-last) for midazolam.
Oral pharmacokinetics (PK) of caffeine after single co-administration with TEV-56286 in healthy volunteers in the fasted state (Part I). | Day 3
  Cmax for caffeine.
Oral pharmacokinetics (PK) of caffeine after single co-administration with TEV-56286 in healthy volunteers in the fasted state (Part I). | Day 3
  PK parameter: AUC(0-inf) for caffeine.
Oral pharmacokinetics (PK) of caffeine after single co-administration with TEV-56286 in healthy volunteers in the fasted state (Part I). | Day 3
  PK parameter: AUC (0-last) for caffeine.
Oral pharmacokinetics (PK) of midazolam after single co-administration with TEV-56286 in healthy volunteers in the fasted state (Part I). | Day 3
  Cmax for midazolam
Oral pharmacokinetics (PK) of midazolam after single co-administration with TEV-56286 in healthy volunteers in the fasted state (Part I). | Day 3
  PK parameter: AUC(0-inf) for midazolam.
Oral pharmacokinetics (PK) of midazolam after single co-administration with TEV-56286 in healthy volunteers in the fasted state (Part I). | Day 3
  PK parameter: AUC (0-last) for midazolam.
Oral pharmacokinetics (PK) of caffeine after repeated administration of TEV-56286 in healthy volunteers in the fasted state (Part I). | Day 18
  PK parameter: Cmax for caffeine.
Oral pharmacokinetics (PK) of caffeine after repeated administration of TEV-56286 in healthy volunteers in the fasted state (Part I). | Day 18
  AUC(0-inf) for caffeine.
Oral pharmacokinetics (PK) of caffeine after repeated administration of TEV-56286 in healthy volunteers in the fasted state (Part I). | Day 18
  PK parameter: AUC (0-last) for caffeine.
Oral pharmacokinetics (PK) of midazolam after repeated administration of TEV-56286 in healthy volunteers in the fasted state (Part I). | Day 18
  PK parameter: Cmax for midazolam.
Oral pharmacokinetics (PK) of midazolam after repeated administration of TEV-56286 in healthy volunteers in the fasted state (Part I). | Day 18
  PK parameter: AUC(0-inf) for midazolam.
Oral pharmacokinetics (PK) of midazolam after repeated administration of TEV-56286 in healthy volunteers in the fasted state (Part I). | Day 18
  PK parameter: AUC (0-last) for midazolam.
Oral pharmacokinetics (PK) of TEV-56286 without fluvoxamine in healthy volunteers after repeated administration in the fasted state (Part II). | Day 14
  PK parameter: Cmax for TEV-56286.
Oral pharmacokinetics (PK) of TEV-56286 without fluvoxamine in healthy volunteers after repeated administration in the fasted state (Part II). | Day 14
  PK parameter: AUC(0-tau) for TEV-56286.
Oral pharmacokinetics (PK) of TEV-56286 in healthy volunteers after repeated co-administration with fluvoxamine in the fasted state. | Day 19
  PK parameter: Cmax for TEV-56286 (Part II).
Oral pharmacokinetics (PK) of TEV-56286 in healthy volunteers after repeated co-administration with fluvoxamine in the fasted state. | Day 19
  PK parameter: AUC(0-tau) for TEV-56286 (Part II).

SECONDARY OUTCOMES:
Oral pharmacokinetics (PK) of substrates caffeine and midazolam | Day 1, Day 3, Day 18
  PK parameter: Tmax
Oral pharmacokinetics (PK) of substrates caffeine and midazolam | Day 1, Day 3, Day 18
  PK parameter: Tlag
Oral pharmacokinetics (PK) of substrates caffeine and midazolam | Day 1, Day 3, Day 18
  PK parameter: lambda-z
Oral pharmacokinetics (PK) of substrates caffeine and midazolam | Day 1, Day 3, Day 18
  PK parameter: T1/2
Oral pharmacokinetics (PK) of substrates caffeine and midazolam | Day 1, Day 3, Day 18
  PK parameter: CL/F
Oral pharmacokinetics (PK) of substrates caffeine and midazolam | Day 1, Day 3, Day 18
  PK parameter: Vz/F
Oral pharmacokinetics (PK) of TEV-56286 after repeated co-administration with fluvoxamine | Day 19
  PK parameter: Tmax
Oral pharmacokinetics (PK) of TEV-56286 after repeated co-administration with fluvoxamine | Day 19
  PK parameter: lambda-z
Oral pharmacokinetics (PK) of TEV-56286 after repeated co-administration with fluvoxamine | Day 19
  PK parameter: T1/2
Oral pharmacokinetics (PK) of TEV-56286 after repeated co-administration with fluvoxamine | Day 19
  PK parameter: CL/F
Oral pharmacokinetics (PK) of TEV-56286 after repeated co-administration with fluvoxamine | Day 19
  PK parameter: Vz/F
Oral pharmacokinetics (PK) of TEV-56286 as perpetrator drug after co-administration with caffeine and midazolam | Day 3
  PK parameter: Tmax
Oral pharmacokinetics (PK) of TEV-56286 as perpetrator drug after co-administration with caffeine and midazolam | Day 3
  PK parameter: Cmax
Oral pharmacokinetics (PK) of TEV-56286 as perpetrator drug after co-administration with caffeine and midazolam | Day 3
  PK parameter: AUC (0-last)
Oral pharmacokinetics (PK) of TEV-56286 | Day 3-18
  PK parameter: Trough concentration for TEV-56286
Oral pharmacokinetics (PK) of TEV-56286 after single co-administration with caffeine and midazolam | Day 18
  PK parameter: Tmax
Oral pharmacokinetics (PK) of TEV-56286 after single co-administration with caffeine and midazolam | Day 18
  PK parameter: Cmax
Oral pharmacokinetics (PK) of TEV-56286 after single co-administration with caffeine and midazolam | Day 18
  PK parameter: Cmin
Oral pharmacokinetics (PK) of TEV-56286 after single co-administration with caffeine and midazolam | Day 18
  PK parameter: Cavg
Oral pharmacokinetics (PK) of TEV-56286 after single co-administration with caffeine and midazolam | Day 18
  PK parameter: AUC (0-tau)
Oral pharmacokinetics (PK) of TEV-56286 after single co-administration with caffeine and midazolam | Day 18
  PK parameter: AUC (0-last)
Oral pharmacokinetics (PK) of fluvoxamine after repeated co-administration with TEV-56286 | Day 19
  PK parameter: Tmax
Oral pharmacokinetics (PK) of fluvoxamine after repeated co-administration with TEV-56286 | Day 19
  PK parameter: Cmax
Oral pharmacokinetics (PK) of fluvoxamine after repeated co-administration with TEV-56286 | Day 19
  PK parameter: Cmin
Oral pharmacokinetics (PK) of fluvoxamine after repeated co-administration with TEV-56286 | Day 19
  PK parameter: Cavg
Oral pharmacokinetics (PK) of fluvoxamine after repeated co-administration with TEV-56286 | Day 19
  PK parameter: AUC (0-tau)
Oral pharmacokinetics (PK) of fluvoxamine after repeated co-administration with TEV-56286 | Day 19
  PK parameter: AUC (0-last)
Oral pharmacokinetics (PK) of fluvoxamine after repeated co-administration with TEV-56286 | Day 15-19
  PK parameter: Trough concentration for fluvoxamine
Oral pharmacokinetics (PK) of TEV-56286 after first dose administered as part of repeated administration | Day 1
  PK parameter: Tlag for TEV-56286
Oral pharmacokinetics (PK) of TEV-56286 following single dose and multiple dose | Day 1, Day 14
  PK parameter: Tmax
Oral pharmacokinetics (PK) of TEV-56286 following single dose and multiple dose | Day 1, Day 14
  PK parameter: Cmax
Oral pharmacokinetics (PK) of TEV-56286 following single dose and multiple dose | Day 1, Day 14
  PK parameter: AUC (0-tau)
Oral pharmacokinetics (PK) of TEV-56286 following single dose and multiple dose | Day 1, Day 14
  PK parameter: lambda-z
Oral pharmacokinetics (PK) of TEV-56286 following single dose and multiple dose | Day 1, Day 14
  PK parameter: T1/2
Oral pharmacokinetics (PK) of TEV-56286 following single dose and multiple dose | Day 1, Day 14
  PK parameter: CL/F
Oral pharmacokinetics (PK) of TEV-56286 following single dose and multiple dose | Day 1, Day 14
  PK parameter: Vz/F
Oral pharmacokinetics (PK) of TEV-56286 following multiple dose | Day 14
  PK parameter: AUC (0-last)
Oral pharmacokinetics (PK) of TEV-56286 following multiple dose | Day 14
  PK parameter: Cmin
Oral pharmacokinetics (PK) of TEV-56286 following multiple dose | Day 14
  PK parameter: Cavg
Oral pharmacokinetics (PK) of TEV-56286 following multiple dose | Day 14
  PK parameter: Accumulation ratio
Oral pharmacokinetics (PK) of metabolites paraxanthine and 1-hydroxy midazolam after single administration of caffeine and midazolam | Day 1, Day 3, Day 18
  PK parameter: Tmax
Oral pharmacokinetics (PK) of metabolites paraxanthine and 1-hydroxy midazolam after single administration of caffeine and midazolam | Day 1, Day 3, Day 18
  PK parameter: Cmax
Oral pharmacokinetics (PK) of metabolites paraxanthine and 1-hydroxy midazolam after single administration of caffeine and midazolam | Day 1, Day 3, Day 18
  PK parameter: AUC (0-last)
Oral pharmacokinetics (PK) of metabolites paraxanthine and 1-hydroxy midazolam after single administration of caffeine and midazolam | Day 1, Day 3, Day 18
  PK parameter: AUC (0-inf)
Oral pharmacokinetics (PK) of metabolites paraxanthine and 1-hydroxy midazolam after single administration of caffeine and midazolam | Day 1, Day 3, Day 18
  PK parameter: lambda-z
Oral pharmacokinetics (PK) of metabolites paraxanthine and 1-hydroxy midazolam after single administration of caffeine and midazolam | Day 1, Day 3, Day 18
  PK parameter: T1/2
Oral pharmacokinetics (PK) of metabolites paraxanthine and 1-hydroxy midazolam after single administration of caffeine and midazolam | Day 1, Day 3, Day 18
  PK parameter: parent: metabolite ratio
Incidence of treatment-emergent adverse events including clinically significant changes in vital signs, ECGs and safety labs | Day 1 up to follow up visit (5-11 days post last TEV-56286 dose)
  adverse events and clinically significant changes in vital signs, ECGs and safety labs
Number of participants reporting use of concomitant medications | Day 1 up to follow up visit (5-11 days post last TEV-56286 dose)
  Number of participants reporting use of concomitant medications
Columbia-Suicide Severity Rating Scale (C-SSRS) total score | Day 3 to day 21
  Columbia-Suicide Severity Rating Scale (C-SSRS) total score

CONTACTS AND LOCATIONS:
Overall Officials: Nand Singh, MD, Principal Investigator — Quotient Sciences Mere Way Ruddington Fields Ruddington Nottingham NG11 6JS, UK
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levin J, Sing N, Melbourne S, Morgan A, Mariner C, Spillantini MG, Wegrzynowicz M, Dalley JW, Langer S, Ryazanov S, Leonov A, Griesinger C, Schmidt F, Weckbecker D, Prager K, Matthias T, Giese A. Safety, tolerability and pharmacokinetics of the oligomer modulator anle138b with exposure levels sufficient for therapeutic efficacy in a murine Parkinson model: A randomised, double-blind, placebo-controlled phase 1a trial. EBioMedicine. 2022 Jun;80:104021. doi: 10.1016/j.ebiom.2022.104021. Epub 2022 Apr 29. PMID 35500536
- [Background] Wagner J, Ryazanov S, Leonov A, Levin J, Shi S, Schmidt F, Prix C, Pan-Montojo F, Bertsch U, Mitteregger-Kretzschmar G, Geissen M, Eiden M, Leidel F, Hirschberger T, Deeg AA, Krauth JJ, Zinth W, Tavan P, Pilger J, Zweckstetter M, Frank T, Bahr M, Weishaupt JH, Uhr M, Urlaub H, Teichmann U, Samwer M, Botzel K, Groschup M, Kretzschmar H, Griesinger C, Giese A. Anle138b: a novel oligomer modulator for disease-modifying therapy of neurodegenerative diseases such as prion and Parkinson's disease. Acta Neuropathol. 2013 Jun;125(6):795-813. doi: 10.1007/s00401-013-1114-9. Epub 2013 Apr 19. PMID 23604588
- [Background] Drug Interaction Studies M12. ICH Harmonised Guideline. International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use. Draft version endorsed on 24 May 2022.
- [Background] Clinical Drug Interaction Studies - Cytochrome P450 Enzyme- and Transporter-Mediated Drug Interactions Guidance for Industry. US Food and Drug Administration. 07 Jul 2020. Available online: https://www.fda.gov/regulatoryinformation/search-fda-guidance-documents/clinical-drug-interaction-studiescytochrome-p450-enzyme-and-transporter-mediated-drug-interactions (accessed 23 Jun 2022).
- See also: Description Sponsor Homepage — http://www.modag.net